CLINICAL TRIAL: NCT01410240
Title: A Prospective, Randomized, Controlled, Single-Blinded, Multicenter Study to Evaluate the Efficacy and Safety of FLOSEAL for Hemostasis in Primary Unilateral Total Knee Arthroplasty (TKA)
Brief Title: Efficacy and Safety of FLOSEAL for Hemostasis in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 611001
Record Dates: First submitted 2011-08-01; First posted 2011-08-05 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-05

CONDITIONS: Knee Replacement Surgery; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Standard of Care; FloSeal Matrix

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (SoC) (Active Comparator): SoC: conventional hemostatic techniques such as cautery and manual compression
  Interventions: Procedure: Standard of Care
- FLOSEAL + Standard of Care (SoC) (Experimental): FLOSEAL: consists of bovine-derived gelatin granules and a human plasma-derived thrombin component.
  SoC: conventional hemostatic techniques such as cautery and manual compression
  Interventions: Drug: FLOSEAL Hemostatic Matrix + Standard of care

INTERVENTIONS:
Procedure: Standard of Care — Conventional hemostatic techniques, such as cautery and manual compression, will be used.
  Arms: Standard of Care (SoC)
Drug: FLOSEAL Hemostatic Matrix + Standard of care — FLOSEAL will be applied topically to areas of the knee where bleeding is observed (e.g. cut bone surfaces, subcutaneous tissue, posterior joint capsule, synovial tissue, medial and lateral gutters, branches of the genicular vessels, and suprapatellar pouch) and will occur intraoperatively. Sufficient amounts of FLOSEAL will be applied quickly using the provided applicators, followed by immediate approximation with a damp gauze, lap pad or sponge for approximately 2 minutes.
  + Standard of care: conventional hemostatic techniques, such as cautery and manual compression, will be used
  Other Names: FLOSEAL
  Arms: FLOSEAL + Standard of Care (SoC)

SUMMARY:
The purpose of this study is to compare the efficacy and safety of FLOSEAL to standard of care for hemostasis in subjects undergoing total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 18 to 80 years of age inclusive at the time of screening
* Participant is planned for primary unilateral total knee arthroplasty
* Participant has signed the informed consent form
* Participant is in stable health (i.e., able to undergo surgery and participate in a follow-up program based on physical examination and medical history)
* Participant has a preoperative Hgb level > 10 g/dL
* If female of childbearing potential, the participant presents with a negative urine pregnancy test and agrees to employ adequate birth control measures for the duration of the study
* Participant is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Participant has had a previous total or partial knee arthroplasty or any surgery on the knee within the previous 6 months
* Participant has osteonecrosis or arthrotomy within the last year
* Participant has prior or current hardware in target knee
* Participant has had injections in the knee:

  1. Steroids within the 3 months prior to scheduled surgery,
  2. Synvisc, Hyalin, etc. within the 6 months prior to scheduled surgery
* Participant has had general surgery within 3 months
* Participant has rheumatoid arthritis or any other inflammatory or traumatic bone injuries to the knee within the 12 months prior to scheduled surgery
* Participant has allergies to products of bovine origin
* Participant has a history of bleeding, platelet, or bone marrow disorders
* Participant has donated more than 1 unit of blood donation in the 3 weeks prior to surgery
* Participant has a history of a coagulation disorder
* Participant is currently taking dipyridamole/ASA (Aggrenox) and/or enoxaparin (Lovenox)
* Participant has been treated with aspirin or Warfarin (Coumadin) or clopidogrel (Plavix) within 7 days prior to surgery
* Participant is not permitted to remain without his/her anti-coagulant regimen (e.g. Plavix) for 48 hours postoperatively
* Participant has taken nonsteroidal anti-inflammatory agents or herbal supplements within 7 days of surgery
* Participant has a history of substance abuse (alcohol, drugs) or is an active smoker
* Participant has liver cirrhosis
* Participant has erythropoietin agonist/stimulating agent within 90 days prior to surgery
* Participant has an active infection or previous history of infection in the affected joint within the previous 6 months
* Participant has participated in another clinical study involving an investigational product (IP) or device within 30 days prior to study enrollment or is scheduled to participate in another clinical study involving an IP or device during the course of this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ildiko Szabo, MD, MBA, Study Director — Baxter Innovations GmbH
Locations (12):
- United States (12):
  - Cedars-Sinai Orthopedic Center, Los Angeles, California
  - Stanford Orthopedics, Redwood City, California
  - Colorado Orthopedic Consultants, PC, Englewood, Colorado
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Florida Research Associates, LLC, DeLand, Florida
  - Shrock Orthopedic Research, LLC, Fort Lauderdale, Florida
  - Phoenix Clinical Research, LLC, Tamarac, Florida
  - Joint Replacement Surgeons of Indiana Foundations, Mooresville, Indiana
  - Rothman Institute, Egg Harbor, New Jersey
  - The Rothman Institute, Philadelphia, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Hill Country Clinical Research, Inc., Austin, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 12 clinical sites in the United States, beginning October 2011
Pre-assignment Details: 137 participants were enrolled and screened. 5 were screen failures. 14 withdrew prior to surgery (1 physician decision, 4 study terminated, 8 withdrawn by participant, 1 sponsor educator not available). 12 were run-in participants. Therefore, 106 of the 137 enrolled were randomized.
Groups:
- FLOSEAL + Standard of Care (SoC): FLOSEAL will be applied topically to areas of the knee where bleeding is observed. FLOSEAL consists of bovine-derived gelatin granules and a human plasma-derived thrombin component.
  SoC: conventional hemostatic techniques such as cautery and manual compression.
- FLOSEAL + Standard of Care (SoC) Run-In Participants: This arm/group only includes the 12 initial "run-in" participants (one for each site permitted to familiarize the investigators with the study procedures and the use of FLOSEAL)
  FLOSEAL will be applied topically to areas of the knee where bleeding is observed. FLOSEAL consists of bovine-derived gelatin granules and a human plasma-derived thrombin component.
  SoC: conventional hemostatic techniques such as cautery and manual compression.
Period: Overall Study
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC) Run-In Participants
Started | 53 | 53 | 12
Completed | 52 | 52 | 10
Not Completed | 1 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Missed week 6 assessments | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- FLOSEAL + Standard of Care (SoC) - Non-Run-In: FLOSEAL will be applied topically to areas of the knee where bleeding is observed. FLOSEAL consists of bovine-derived gelatin granules and a human plasma-derived thrombin component.
  Standard of Care: Conventional hemostatic techniques, such as cautery and manual compression
- FLOSEAL + Standard of Care (SoC) - Run-In: Run-In = The first participant who qualified for surgery at each site was treated with FLOSEAL + SoC to allow the investigator to familiarize with the study procedures and the use of FLOSEAL.
  FLOSEAL will be applied topically to areas of the knee where bleeding is observed. FLOSEAL consists of bovine-derived gelatin granules and a human plasma-derived thrombin component.
  Standard of Care: Conventional hemostatic techniques, such as cautery and manual compression
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC) - Non-Run-In | FLOSEAL + Standard of Care (SoC) - Run-In | Total
Number analyzed (Participants) | 53 | 53 | 12 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (8.09) | 64.8 (7.73) | 59.4 (8.49) | 64.8 (8.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 7 | 65
  Male | 24 | 24 | 5 | 53
Region of Enrollment [Number; unit: participants]
  United States | 53 | 53 | 12 | 118

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin (Hgb) Level at Day 2 Post-operatively
Time Frame: Pre-operative and 2 days post-operatively
Population: Full Analysis Set
  Participants who required a transfusion prior to the primary outcome assessment of Hgb level at postoperative Day 2 were excluded from the primary outcome analysis.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 46 | 41
g/dL | -3.73 (1.497) | -3.70 (1.205)
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Test type: Superiority or Other; p = 0.453, one-sided, two-sample t-test

2. Secondary Outcome: Change in Hemoglobin (Hgb) Levels at Day 1 Post-operatively
Time Frame: Pre-operative and day 1 post-operatively
Population: Full Analysis Set
  Participants who required a transfusion prior to the outcome assessments were excluded from the efficacy analyses of Hgb levels.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 48 | 45
g/dL | -3.02 (1.069) | -3.15 (1.217)
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Test type: Superiority or Other; p = 0.708, one-sided, two-sample t-test

3. Secondary Outcome: Change in Hemoglobin (Hgb) Levels at Day 3 Post-operatively
Description: Participants who required a transfusion prior to the outcome assessments were excluded from the efficacy analyses of Hgb levels.
Time Frame: Pre-operative and day 3 post-operatively
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 39 | 31
g/dL | -3.81 (1.427) | -3.84 (1.324)
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Test type: Superiority or Other; p = 0.527, one-sided, two-sample t-test

4. Secondary Outcome: Change From Baseline in Hematocrit (Hct) at Postoperative Day 1
Description: Participants who required a transfusion prior to the outcome assessments were excluded from the efficacy analyses of Hct levels.
Time Frame: Pre-operative and day 1 post-operatively
Population: Full Analysis Set
  Participants who required a transfusion prior to the outcome assessments were excluded from the efficacy analyses of Hct levels.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 48 | 45
percent | -9.0 (3.85) | -8.8 (3.92)
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Test type: Superiority or Other; p = 0.561, one-sided Wilcoxon rank sum test

5. Secondary Outcome: Change From Baseline in Hematocrit (Hct) at Postoperative Day 2
Time Frame: Pre-operative and day 2 post-operatively
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 44 | 40
percent | -11.2 (4.67) | -10.6 (4.21)
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Test type: Superiority or Other; p = 0.356, one-sided Wilcoxon rank sum test

6. Secondary Outcome: Change From Baseline in Hematocrit (Hct) at Postoperative Day 3
Time Frame: Pre-operative and day 3 post-operatively
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 39 | 31
percent | -11.1 (4.46) | -11.0 (4.31)
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Test type: Superiority or Other; p = 0.533, one-sided Wilcoxon rank sum test

7. Secondary Outcome: Total Tourniquet Time
Description: Measured from the time point of the tourniquet inflation to deflation using the same watch/clock
Time Frame: Intra-operatively (on day of surgery = Day 0)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 50 | 47
minutes | 49.2 (19.76) | 47.3 (17.45)
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Test type: Superiority or Other; p = 0.734, two-sided Wilcoxon rank sum test

8. Secondary Outcome: Amount of FLOSEAL Applied
Time Frame: Intra-operatively (Day 0)
Population: Safety Analysis Set
  Note: The FLOSEAL (+ Standard of Care (SoC)) Arm/Group Includes the 15 Run-In participants
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 65
mL | 18.1 (5.52)

9. Secondary Outcome: Duration of Surgery
Time Frame: Time from first incision to complete wound closure (Day 0)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 50 | 47
minutes | 74.5 (19.73) | 76.9 (17.33)

10. Secondary Outcome: Transfusion Requirements - Packed Red Blood Cells
Time Frame: Intra-operatively (Day 0) thru Postoperative Day 3
Population: Full Analysis Set - participants with transfusion requirement
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 10 | 12
mL | 484.0 (173.54) | 403.3 (157.90)
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Test type: Superiority or Other; p = 0.314, two-sided Wilcoxon rank sum test

11. Secondary Outcome: Total Drain Output at Day 1 Post-operatively
Time Frame: 1 day post-operatively
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 49 | 47
mL | 839.6 (476.38) | 647.3 (338.96)
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Test type: Superiority or Other; p = 0.063, two-sided Wilcoxon rank sum test

12. Secondary Outcome: Pain Management - Number of Days When Pain Medication Was Used
Description: Each participant kept a knee pain management diary. The diary was used to document the pain medication taken on a daily basis.
  While the participants were hospitalized, either they filled out the diary, or study team members collected the pain diary data and filled out the diary.
Time Frame: Pre-operatively (Day -1 to Day 0); and post-operatively daily thru week 6
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 50 | 47
days
  All pain medications | 28.7 (13.71) | 31.9 (12.72)
  Narcotics | 25.1 (13.66) | 30.3 (12.84)

13. Secondary Outcome: Visual Analogue Scale (VAS) Pain Scores
Description: Participant rated assessment of the level of pain they are experiencing with their operated knee. The VAS Pain Scale rates pain on a scale from 0 (no pain) to 10 (worst possible pain). For the pain scale, a higher score indicates worse pain.
Time Frame: Pre-operatively (Day -1 to Day 0) and post-operatively at Day 3, Week 1, 2 and 6
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 50 | 47
score on a scale
  Baseline (N= 50, 47) | 4.9 (3.03) | 4.4 (2.76)
  Day 3 Postoperative (N= 45, 42) | 3.2 (2.60) | 4.1 (2.43)
  Week 1 Postoperative (N= 40, 40) | 4.4 (2.13) | 4.8 (2.08)
  Week 2 Postoperative (N= 40, 42) | 3.0 (1.87) | 3.8 (2.12)
  Week 6 Postoperative (N= 49, 46) | 1.3 (1.34) | 2.4 (1.86)

14. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Pain Scores at Postoperative Day 3
Description: as for outcome 13
Time Frame: Pre-operatively (Day -1 to Day 0) and post-operatively at Day 3
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 45 | 42
score on a scale | -1.6 (3.18) | -0.1 (3.54)
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Test type: Superiority or Other; p = 0.058, two-sided Wilcoxon rank sum test

15. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Pain Scores at Postoperative Week 1
Description: as for outcome 13
Time Frame: Pre-operatively (Day -1 to Day 0) and post-operatively at Week 1
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 40 | 40
score on a scale | -0.4 (2.88) | 0.4 (2.97)
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Test type: Superiority or Other; p = 0.421, two-sided Wilcoxon rank sum test

16. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Pain Scores at Postoperative Week 2
Description: as for outcome 13
Time Frame: Pre-operatively (Day -1 to Day 0) and post-operatively at Week 2
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 40 | 42
score on a scale | -1.8 (2.64) | -0.5 (3.18)
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Test type: Superiority or Other; p = 0.161, two-sided Wilcoxon rank sum test

17. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Pain Scores at Postoperative Week 6
Description: as for outcome 13
Time Frame: Pre-operatively (Day -1 to Day 0) and post-operatively at Week 6
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 49 | 46
score on a scale | -3.5 (2.65) | -2.1 (2.52)
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Test type: Superiority or Other; p = 0.016, two-sided Wilcoxon rank sum test

18. Secondary Outcome: Western Ontario and McMaster Universities (WOMAC) Function Index Scores
Description: A well-validated scale to reflect problems in people with lower limb issues.
  1. Pain scale (5 items): 0 (none) to 10 (extreme pain) is used to grade each item, higher scores indicate greater pain. The overall pain scale = 0 (no pain) to 50 (extreme pain)
  2. Stiffness scale (2 items): 0 (none) to 10 (extreme stiffness) is used to grade each item, higher scores indicate greater stiffness. The overall stiffness scale = 0 (no stiffness) to 20 (extreme stiffness)
  3. Physical Activity Difficulty (PAD) scale (17 items): 0 (none) to 10 (extreme PAD) is used to grade each item, with higher scores indicating greater PAD. The overall PAD scale = 0 (no PAD) to 170 (extreme PAD)
  Averages calculated by taking sum of all individual item scores listed above and dividing by total number of items, range = 0 (no issues) to 10 (extreme issues).
  Total Scores calculated by taking sum of all individual item scores listed above, range = 0 (no issues) to 240 (extreme issues)
  Postoperative (Postop)
Time Frame: Pre-operatively (Day -1 to Day 0), and post-operatively at Day 3 and Week 1, 2 and 6
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 50 | 47
score on a scale
  Baseline: Pain (N= 50, 47) | 26.8 (11.81) | 27.6 (10.69)
  Baseline: Stiffness (N= 50, 47) | 11.9 (4.86) | 11.6 (5.31)
  Baseline: Physical Functioning (N= 47, 43) | 91.3 (37.75) | 92.3 (34.51)
  Baseline: Average (N= 47, 43) | 5.4 (2.18) | 5.5 (1.97)
  Baseline: Total Score (N= 47, 43) | 129.7 (52.27) | 130.9 (47.36)
  Day 3 Postoperative: Pain (N= 46, 42) | 19.1 (11.87) | 21.5 (10.28)
  Day 3 Postoperative: Stiffness (N= 46, 42) | 10.2 (4.64) | 11.1 (3.37)
  Day 3 Post-op: Physical Functioning (N= 15, 16) | 91.7 (37.90) | 97.8 (37.85)
  Day 3 Post-op: Average (N= 15, 16) | 5.2 (2.12) | 5.6 (2.05)
  Day 3 Post-op: Total Score (N= 15, 16) | 124.7 (50.99) | 133.9 (49.17)
  Week 1 Post-op: Pain (N= 41, 41) | 23.5 (11.54) | 24.5 (11.25)
  Week 1 Post-op: Stiffness (N= 41, 40) | 11.8 (4.57) | 12.2 (4.48)
  Week 1 Post-op: Physical Functioning (N= 18, 24) | 77.0 (37.77) | 76.7 (41.11)
  Week 1 Post-op: Average (N= 18, 24) | 4.7 (2.18) | 4.7 (2.19)
  Week 1 Post-op: Total Score (N= 18, 24) | 112.3 (52.42) | 112.3 (52.66)
  Week 2 Post-op: Pain (N= 41, 43) | 15.4 (8.07) | 19.9 (11.04)
  Week 2 Post-op: Stiffness (N= 41, 42) | 8.1 (4.00) | 10.2 (4.07)
  Week 2 Post-op: Physical Functioning (N= 26, 28) | 51.3 (25.74) | 68.5 (37.20)
  Week 2 Post-op: Average (N= 25, 28) | 3.0 (1.39) | 4.1 (2.09)
  Week 2 Post-op: Total Score (N= 25, 28) | 72.5 (33.24) | 99.6 (50.09)
  Week 6 Post-op: Pain (N= 49, 47) | 8.5 (7.60) | 12.6 (7.98)
  Week 6 Post-op: Stiffness (N= 49, 46) | 5.5 (3.64) | 7.7 (3.96)
  Week 6 Post-op: Physical Functioning (N= 43, 43) | 27.5 (25.78) | 39.9 (26.98)
  Week 6 Post-op: Average (N= 43, 42) | 1.7 (1.51) | 2.5 (1.52)
  Week 6 Post-op: Total Score (N= 43, 42) | 41.6 (36.24) | 61.1 (36.56)

19. Secondary Outcome: Change From Baseline at Postoperative Day 3, Week 1, Week 2, and Week 6 in Western Ontario and McMaster Universities (WOMAC) Scores
Description: A well-validated scale to reflect problems in people with lower limb issues.
  1. Pain scale (5 items): 0 (none) to 10 (extreme pain) is used to grade each item, higher scores indicate greater pain. The overall pain scale = 0 (no pain) to 50 (extreme pain)
  2. Stiffness scale (2 items): 0 (none) to 10 (extreme stiffness) is used to grade each item, higher scores indicate greater stiffness. The overall stiffness scale = 0 (no stiffness) to 20 (extreme stiffness)
  3. Physical Activity Difficulty (PAD) scale (17 items): 0 (none) to 10 (extreme PAD) is used to grade each item, with higher scores indicating greater PAD. The overall PAD scale = 0 (no PAD) to 170 (extreme PAD) Averages calculated by taking sum of all individual item scores listed above and dividing by total number of items, range = 0 (no issues) to 10 (extreme issues).
  Total Scores calculated by taking sum of all individual item scores listed above, range = 0 (no issues) to 240 (extreme issues).
  Postoperative (Postop)
Time Frame: Pre-operatively (Day -1 to Day 0), and post-operatively at Day 3 and Week 1, 2 and 6
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 49 | 47
score on a scale
  Change Day 3: Pain (N= 46, 42) | -7.3 (12.72) | -5.1 (12.43)
  Change Day 3: Stiffness (N= 46, 42) | -1.7 (5.79) | -0.1 (4.90)
  Change Day 3: Physical Functioning (N= 15, 16) | 4.7 (39.93) | 17.0 (39.37)
  Change Day 3: Average (N= 15, 16) | -0.0 (2.15) | 0.8 (2.28)
  Change Day 3: Total Score (N= 15, 16) | 0.0 (51.66) | 19.2 (54.70)
  Change Week 1: Pain (N= 41, 41) | -3.2 (11.54) | -3.2 (10.23)
  Change Week 1: Stiffness (N= 41, 40) | -0.2 (6.36) | 0.5 (6.05)
  Change Week 1: Physical Functioning (N= 18, 24) | -16.7 (42.58) | -7.3 (44.39)
  Change Week 1: Average (N= 18, 24) | -0.9 (2.38) | -0.3 (2.28)
  Change Week 1: Total Score (N= 18, 24) | -22.0 (57.04) | -6.2 (54.60)
  Change Week 2: Pain (N= 41, 43) | -11.2 (10.90) | -7.8 (11.98)
  Change Week 2: Stiffness (N= 41, 42) | -3.8 (5.84) | -1.7 (6.39)
  Change Week 2: Physical Functioning (N= 26, 28) | -40.3 (33.65) | -18.7 (43.74)
  Change Week 2: Average (N= 25, 28) | -2.3 (1.95) | -1.0 (2.39)
  Change Week 2: Total Score (N= 25, 28) | -55.5 (46.91) | -24.5 (57.34)
  Change Week 6: Pain (N= 49, 47) | -18.3 (10.46) | -15.0 (12.10)
  Change Week 6: Stiffness (N= 49, 46) | -6.5 (5.54) | -4.0 (6.34)
  Change Week 6: Physical Functioning (N= 42, 40) | -63.6 (38.27) | -48.9 (33.69)
  Change Week 6: Average (N= 42, 39) | -3.6 (2.16) | -2.8 (1.95)
  Change Week 6: Total Score (N= 42, 39) | -87.0 (51.80) | -66.5 (46.90)
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Day 3: Pain; Test type: Superiority or Other; p = 0.534, two-sided Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Day 3: Stiffness; Test type: Superiority or Other; p = 0.269, two-sided Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Day 3: Physical Functioning; Test type: Superiority or Other; p = 0.693, two-sided Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Day 3: Average Score; Test type: Superiority or Other; p = 0.343, two-sided Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Day 3: Total Score; Test type: Superiority or Other; p = 0.343, two-sided Wilcoxon rank sum test
Statistical Analysis 6: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 1: Pain; Test type: Superiority or Other; p = 0.978, two-sided Wilcoxon rank sum test
Statistical Analysis 7: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 1: Stiffness; Test type: Superiority or Other; p = 0.709, two-sided Wilcoxon rank sum test
Statistical Analysis 8: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 1: Physical Functioning; Test type: Superiority or Other; p = 0.594, two-sided Wilcoxon rank sum test
Statistical Analysis 9: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 1: Average Score; Test type: Superiority or Other; p = 0.501, two-sided Wilcoxon rank sum test
Statistical Analysis 10: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 1: Total Score; Test type: Superiority or Other; p = 0.501, two-sided Wilcoxon rank sum test
Statistical Analysis 11: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 2: Pain; Test type: Superiority or Other; p = 0.171, two-sided Wilcoxon rank sum test
Statistical Analysis 12: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 2: Stiffness; Test type: Superiority or Other; p = 0.077, two-sided Wilcoxon rank sum test
Statistical Analysis 13: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 2: Physical Functioning; Test type: Superiority or Other; p = 0.026, two-sided Wilcoxon rank sum test
Statistical Analysis 14: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 2: Average Score; Test type: Superiority or Other; p = 0.012, two-sided Wilcoxon rank sum test
Statistical Analysis 15: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 2: Total Score; Test type: Superiority or Other; p = 0.012, two-sided Wilcoxon rank sum test
Statistical Analysis 16: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 6: Pain; Test type: Superiority or Other; p = 0.126, two-sided Wilcoxon rank sum test
Statistical Analysis 17: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 6: Stiffness; Test type: Superiority or Other; p = 0.044, two-sided Wilcoxon rank sum test
Statistical Analysis 18: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Test type: Superiority or Other; p = 0.153, two-sided Wilcoxon rank sum test — Change Week 6: Physical Functioning
Statistical Analysis 19: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 6: Average Score; Test type: Superiority or Other; p = 0.134, two-sided Wilcoxon rank sum test
Statistical Analysis 20: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 6: Total Score; Test type: Superiority or Other; p = 0.134, two-sided Wilcoxon rank sum test

20. Secondary Outcome: Quality of Life (Utilizing the Short Form 36 Health Survey [SF-36]) Measured Preoperatively (Baseline), and Postoperatively at Week 1, 2, and 6
Description: Physical Functioning (PF); Role Limitation Due to Physical Health (RP); Bodily Pain (BP); General Health (GH); Vitality (VT); Social Functioning (SF); Role Limitation Due to Emotional Problems (RE); Mental Health (MH), Physical Component Score (PCS); Mental Component Score (MCS). Scores range 0-100, higher scores represent better health. There is no total overall score; scoring is done for subscores and summary scores. Scores were included where data was available.
Time Frame: Preoperative, and Postoperative Weeks 1, 2, and 6
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 50 | 47
Scores on a scale
  Baseline PF (N= 49, 47) | 24.9 (6.37) | 25.8 (7.81)
  Baseline RP (N= 50, 47) | 32.9 (10.87) | 33.5 (11.06)
  Baseline BP (N= 50, 47) | 35.5 (7.58) | 36.2 (9.21)
  Baseline GH (N= 49, 47) | 52.3 (6.34) | 50.2 (9.83)
  Baseline VT (N= 49, 47) | 47.9 (10.73) | 47.3 (9.98)
  Baseline SF (N= 50, 47) | 42.1 (11.73) | 44.9 (12.18)
  Baseline RE (N= 49, 47) | 40.7 (14.11) | 45.8 (14.29)
  Baseline MH (N= 49, 47) | 48.9 (10.25) | 50.2 (10.32)
  Baseline PCS (N= 48, 47) | 31.4 (7.11) | 30.3 (8.41)
  Baseline MCS (N= 48, 47) | 52.3 (12.46) | 55.2 (12.28)
  Change Week 1: PF (N= 39, 37) | 23.1 (7.88) | 22.9 (8.16)
  Change Week 1: RP (N= 38, 37) | 25.3 (8.02) | 26.5 (9.99)
  Change Week 1: BP (N= 40, 40) | 33.9 (7.99) | 33.1 (8.09)
  Change Week 1: GH (N= 41, 40) | 52.9 (5.43) | 50.1 (10.09)
  Change Week 1: VT (N= 40, 40) | 43.3 (11.02) | 42.0 (10.64)
  Change Week 1: SF (N= 40, 40) | 33.0 (12.70) | 37.1 (14.12)
  Change Week 1: RE (N= 37, 38) | 36.8 (17.03) | 39.5 (17.97)
  Change Week 1: MH (N= 40, 40) | 48.0 (10.35) | 50.0 (9.96)
  Change Week 1: PCS (N= 36, 37) | 28.4 (7.26) | 26.6 (7.16)
  Change Week 1: MCS (N= 36, 37) | 47.9 (12.38) | 51.1 (13.18)
  Change Week 2: PF (N= 40, 38) | 26.0 (8.40) | 24.3 (7.06)
  Change Week 2: RP (N= 36, 42) | 28.1 (9.47) | 26.7 (7.35)
  Change Week 2: BP (N= 40, 42) | 38.8 (7.34) | 35.1 (6.01)
  Change Week 2: GH (N= 40, 42) | 52.4 (6.91) | 51.9 (9.59)
  Change Week 2: VT (N= 40, 42) | 47.6 (6.55) | 45.8 (10.60)
  Change Week 2: SF (N= 40, 42) | 39.4 (9.50) | 37.6 (12.82)
  Change Week 2: RE (N= 35, 41) | 38.9 (15.81) | 40.2 (15.97)
  Change Week 2: MH (N= 40, 42) | 50.7 (10.18) | 51.5 (10.32)
  Change Week 2: PCS (N= 33, 37) | 30.5 (7.72) | 27.8 (7.33)
  Change Week 2: MCS (N= 33, 37) | 51.7 (13.00) | 53.2 (10.89)
  Change Week 6: PF (N= 47, 46) | 37.0 (11.13) | 34.0 (9.75)
  Change Week 6: RP (N= 49, 47) | 41.8 (11.05) | 38.8 (11.03)
  Change Week 6: BP (N= 49, 47) | 47.7 (9.20) | 43.9 (8.43)
  Change Week 6: GH (N= 49, 47) | 54.2 (6.41) | 52.7 (9.44)
  Change Week 6: VT (N= 49, 47) | 53.4 (10.31) | 49.1 (9.63)
  Change Week 6: SF (N= 49, 47) | 48.2 (10.50) | 47.3 (10.94)
  Change Week 6: RE (N= 49, 47) | 46.5 (12.52) | 46.5 (12.57)
  Change Week 6: MH (N= 49, 47) | 54.0 (8.96) | 52.3 (11.24)
  Change Week 6: PCS (N= 47, 46) | 41.7 (8.87) | 38.1 (9.29)
  Change Week 6: MCS (N= 47, 46) | 54.5 (8.96) | 55.1 (11.32)

21. Secondary Outcome: Change From Baseline in SF-36 Scores at Postoperative Weeks 1, 2, and 6
Description: Physical Functioning (PF); Role Limitation Due to Physical Health (RP); Bodily Pain (BP); General Health (GH); Vitality (VT); Social Functioning (SF); Role Limitation Due to Emotional Problems (RE); Mental Health (MH), Physical Component Score (PCS); Mental Component Score (MCS). Scores range 0-100, higher scores represent better health. There is no total overall score; scoring is done for subscores and summary scores. Scores were included where data was available.
  Change in SF-36 Scores From Baseline = (Postoperative Week 1,2, or 6 Scores) - (Baseline Scores).
Time Frame: Baseline and Postoperative Weeks 1, 2, and 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 50 | 47
Scores on a scale
  Change Week 1: PF (N= 38, 37) | -2.1 (10.18) | -2.7 (9.09)
  Change Week 1: RP (N= 38, 37) | -8.0 (10.05) | -6.6 (11.39)
  Change Week 1: BP (N= 40, 40) | -2.3 (10.93) | -3.4 (9.65)
  Change Week 1: GH (N= 40, 40) | 0.1 (6.23) | -1.1 (7.68)
  Change Week 1: VT (N= 39, 40) | -5.9 (9.66) | -5.7 (11.81)
  Change Week 1: SF (N= 40, 40) | -10.8 (12.75) | -6.7 (15.30)
  Change Week 1: RE (N= 36, 38) | -3.9 (16.85) | -6.2 (20.12)
  Change Week 1: MH (N= 39, 40) | -2.3 (10.79) | -0.4 (11.26)
  Change Week 1: PCS (N= 34, 37) | -3.8 (8.97) | -3.5 (7.73)
  Change Week 1: MCS (N= 34, 37) | -5.1 (10.60) | -4.1 (14.13)
  Change Week 2: PF (N= 39, 38) | 1.1 (10.21) | -1.2 (7.07)
  Change Week 2: RP (N= 36, 42) | -4.6 (12.48) | -6.9 (9.08)
  Change Week 2: BP (N= 40, 42) | 2.8 (7.90) | -1.4 (9.39)
  Change Week 2: GH (N= 39, 42) | -0.0 (6.26) | 1.0 (8.92)
  Change Week 2: VT (N= 39, 42) | -0.5 (9.07) | -2.1 (12.39)
  Change Week 2: SF (N= 40, 42) | -3.5 (10.95) | -6.4 (13.14)
  Change Week 2: RE (N= 34, 41) | -0.7 (16.89) | -6.6 (16.08)
  Change Week 2: MH (N= 39, 42) | 0.8 (12.36) | 0.5 (12.83)
  Change Week 2: PCS (N= 32, 37) | -0.9 (7.76) | -2.4 (6.89)
  Change Week 2: MCS (N= 32, 37) | 0.3 (12.90) | -2.0 (12.83)
  Change Week 6: PF (N= 46, 46) | 12.0 (11.34) | 8.0 (7.89)
  Change Week 6: RP (N= 49, 47) | 8.7 (14.84) | 5.4 (12.20)
  Change Week 6: BP (N= 49, 47) | 12.3 (10.43) | 7.7 (10.00)
  Change Week 6: GH (N= 48, 47) | 1.9 (6.33) | 2.5 (9.73)
  Change Week 6: VT (N= 48, 47) | 5.7 (15.00) | 1.8 (11.95)
  Change Week 6: SF (N= 49, 47) | 5.8 (14.62) | 2.4 (13.64)
  Change Week 6: RE (N= 48, 47) | 5.9 (17.20) | 0.7 (14.76)
  Change Week 6: MH (N= 48, 47) | 5.2 (11.90) | 2.1 (14.52)
  Change Week 6: PCS (N= 45, 46) | 10.4 (10.43) | 7.8 (8.62)
  Change Week 6: MCS (N= 45, 46) | 2.1 (12.53) | -0.2 (13.97)
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 1: Physical Functioning; Test type: Superiority or Other; p = 0.962, two-sided Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 1: Role-Physical; Test type: Superiority or Other; p = 0.714, two-sided Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 1: Bodily Pain; Test type: Superiority or Other; p = 0.668, two-sided Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 1: General Health; Test type: Superiority or Other; p = 0.556, two-sided Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 1: Vitality; Test type: Superiority or Other; p = 0.705, two-sided Wilcoxon rank sum test
Statistical Analysis 6: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 1: Social Functioning; Test type: Superiority or Other; p = 0.122, two-sided Wilcoxon rank sum test
Statistical Analysis 7: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 1: Role-Emotional; Test type: Superiority or Other; p = 0.254, two-sided Wilcoxon rank sum test
Statistical Analysis 8: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 1: Mental Health; Test type: Superiority or Other; p = 0.500, two-sided Wilcoxon rank sum test
Statistical Analysis 9: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 1: Physical Component Summary; Test type: Superiority or Other; p = 0.849, two-sided Wilcoxon rank sum test
Statistical Analysis 10: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 1: Mental Component Summary; Test type: Superiority or Other; p = 0.959, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 2: Physical Functioning; Test type: Superiority or Other; p = 0.574, two-sided Wilcoxon rank sum test
Statistical Analysis 12: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 2: Role-Physical; Test type: Superiority or Other; p = 0.524, two-sided Wilcoxon rank sum test
Statistical Analysis 13: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 2: Bodily Pain; Test type: Superiority or Other; p = 0.049, two-sided Wilcoxon rank sum test
Statistical Analysis 14: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 2: General Health; Test type: Superiority or Other; p = 0.447, two-sided Wilcoxon rank sum test
Statistical Analysis 15: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 2: Vitality; Test type: Superiority or Other; p = 0.823, two-sided Wilcoxon rank sum test
Statistical Analysis 16: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 2: Social Functioning; Test type: Superiority or Other; p = 0.661, two-sided Wilcoxon rank sum test
Statistical Analysis 17: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 2: Role-Emotional; Test type: Superiority or Other; p = 0.086, two-sided Wilcoxon rank sum test
Statistical Analysis 18: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 2: Mental Health; Test type: Superiority or Other; p = 0.635, two-sided Wilcoxon rank sum test
Statistical Analysis 19: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 2: Physical Component Summary; Test type: Superiority or Other; p = 0.481, two-sided Wilcoxon rank sum test
Statistical Analysis 20: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 2: Mental Component Summary; Test type: Superiority or Other; p = 0.140, two-sided Wilcoxon rank sum test
Statistical Analysis 21: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 6: Physical Functioning; Test type: Superiority or Other; p = 0.107, two-sided Wilcoxon rank sum test
Statistical Analysis 22: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 6: Role-Physical; Test type: Superiority or Other; p = 0.298, two-sided Wilcoxon rank sum test
Statistical Analysis 23: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 6: Bodily Pain; Test type: Superiority or Other; p = 0.071, two-sided Wilcoxon rank sum test
Statistical Analysis 24: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 6: General Health; Test type: Superiority or Other; p = 0.940, two-sided Wilcoxon rank sum test
Statistical Analysis 25: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 6: Vitality; Test type: Superiority or Other; p = 0.293, two-sided Wilcoxon rank sum test
Statistical Analysis 26: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 6: Social Functioning; Test type: Superiority or Other; p = 0.265, two-sided Wilcoxon rank sum test
Statistical Analysis 27: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 6: Role-Emotional; Test type: Superiority or Other; p = 0.036, two-sided Wilcoxon rank sum test
Statistical Analysis 28: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 6: Mental Health; Test type: Superiority or Other; p = 0.307, two-sided Wilcoxon rank sum test
Statistical Analysis 29: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 6: Physical Component Summary; Test type: Superiority or Other; p = 0.448, two-sided Wilcoxon rank sum test
Statistical Analysis 30: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Change Week 6: Mental Component Summary; Test type: Superiority or Other; p = 0.255, two-sided Wilcoxon rank sum test

22. Primary Outcome: Proportion of Participants Who Have Adverse Events Related to Investigational Product (IP)
Description: * Proportion of Participants who have serious injuries (SIs) related to IP
  * Proportion of Participants who have non-serious adverse events (non-SAEs) related to IP
Time Frame: Throughout the study period, 1 year and 4 months
Population: Safety Analysis Set
  Note: The FLOSEAL (+ Standard of Care (SoC)) Arm/Group Includes the 12 Run-In participants
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | FLOSEAL + Standard of Care (SoC) | Standard of Care (SoC)
Number analyzed (Participants) | 65 | 53
Proportion of participants
  Participants who have SIs related to IP | 0.00 [0.000 to 0.055] | 0.00 [0.000 to 0.067]
  Participants who have non-SAEs related to IP | 0.02 [0.000 to 0.083] | 0.00 [0.000 to 0.067]

23. Secondary Outcome: Length of Hospital Stay
Time Frame: From the day of hospitalization to the day of discharge
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Standard of Care (SoC) | FLOSEAL + Standard of Care (SoC)
Number analyzed (Participants) | 50 | 47
Days | 3.52 (0.857) | 3.38 (0.918)
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs FLOSEAL + Standard of Care (SoC); Test type: Superiority or Other; p = 0.052, two-sided Wilcoxon rank sum test

24. Secondary Outcome: Proportion of Participants With Transfusion Requirements
Time Frame: Intra-operative
Population: Safety Analysis Set
  Note: The FLOSEAL (+ Standard of Care (SoC)) Arm/Group Includes the 12 Run-In participants
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Groups:
- FLOSEAL + Standard of Care (SoC) Including Run-In Participants: FLOSEAL will be applied topically to areas of the knee where bleeding is observed. FLOSEAL consists of bovine-derived gelatin granules and a human plasma-derived thrombin component.
  SoC: conventional hemostatic techniques such as cautery and manual compression.
  Run-In = The first participant who qualified for surgery at each site was treated with FLOSEAL + SoC to allow the investigator to familiarize with the study procedures and the use of FLOSEAL.
Arm/Group | FLOSEAL + Standard of Care (SoC) Including Run-In Participants | Standard of Care (SoC)
Number analyzed (Participants) | 65 | 53
Proportion of participants | 0.25 [0.148 to 0.369] | 0.19 [0.094 to 0.320]

25. Secondary Outcome: Proportion of Participants With Wound Complications (ie, Hematoma, Cellulitis, Dehiscence, Superficial or Deep Infection, and Persistent Drainage)
Time Frame: Day 0; Post-operative Days 1, 3 and Weeks 1, 2, 6
Population: Safety Analysis Set
  Note: The FLOSEAL (+ Standard of Care (SoC)) Arm/Group Includes the 12 Run-In participants
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | FLOSEAL + Standard of Care (SoC) Including Run-In Participants | Standard of Care (SoC)
Number analyzed (Participants) | 65 | 53
Proportion of participants | 0.03 [0.004 to 0.107] | 0.06 [0.012 to 0.157]

26. Secondary Outcome: Proportion of Participants With Any Adverse Events or Serious Injuries During or After Surgery
Time Frame: Day 0; Post-operative Days 1, 3 and Weeks 1, 2, 6
Population: Safety Analysis Set
  Note: The FLOSEAL (+ Standard of Care (SoC)) Arm/Group Includes the 12 Run-In participants
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | FLOSEAL + Standard of Care (SoC) Including Run-In Participants | Standard of Care (SoC)
Number analyzed (Participants) | 65 | 53
Proportion of participants | 0.26 [0.160 to 0.385] | 0.36 [0.231 to 0.502]

27. Secondary Outcome: Rehabilitation Parameter by Study Day- Number of Participants Who Saw Their Physical Therapist
Description: The number of participants responding affirmative in their rehabilitation diaries for each day
Time Frame: 60 days
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | FLOSEAL + Standard of Care (SoC) | Standard of Care (SoC)
Number analyzed (Participants) | 45 | 49
participants
  Day 1 (N= 45, 48) | 24 | 22
  Day 2 (N= 45, 49) | 42 | 47
  Day 3 (N= 44, 49) | 43 | 48
  Day 4 (N= 45, 47) | 41 | 46
  Day 5 (N= 39, 42) | 27 | 31
  Day 6 (N= 35, 39) | 17 | 16
  Day 7 (N= 37, 39) | 20 | 18
  Day 8 (N= 37, 42) | 19 | 24
  Day 9 (N= 35, 39) | 13 | 19
  Day 10 (N= 32, 38) | 17 | 20
  Day 11 (N= 35, 41) | 12 | 21
  Day 12 (N= 34, 37) | 10 | 19
  Day 13 (N= 36, 38) | 14 | 13
  Day 14 (N= 39, 36) | 15 | 15
  Day 15 (N= 39, 41) | 21 | 24
  Day 16 (N= 39, 41) | 16 | 20
  Day 17 (N= 37, 41) | 20 | 21
  Day 18 (N= 38, 41) | 13 | 21
  Day 19 (N= 40, 40) | 18 | 15
  Day 20 (N= 38, 40) | 4 | 9
  Day 21 (N= 38, 40) | 16 | 10
  Day 22 (N= 38, 41) | 12 | 14
  Day 23 (N= 38, 39) | 14 | 10
  Day 24 (N= 39, 39) | 8 | 12
  Day 25 (N= 37, 40) | 9 | 13
  Day 26 (N= 38, 39) | 8 | 9
  Day 27 (N= 38, 38) | 3 | 2
  Day 28 (N= 37, 39) | 9 | 8
  Day 29 (N= 38, 39) | 15 | 13
  Day 30 (N= 36, 40) | 10 | 17
  Day 31 (N= 35, 40) | 7 | 10
  Day 32 (N= 37, 40) | 13 | 14
  Day 33 (N= 37, 39) | 8 | 13
  Day 34 (N= 37, 39) | 7 | 6
  Day 35 (N= 38, 39) | 13 | 6
  Day 36 (N= 38, 39) | 15 | 13
  Day 37 (N= 35, 38) | 10 | 10
  Day 38 (N= 35, 41) | 9 | 12
  Day 39 (N= 36, 39) | 11 | 15
  Day 40 (N= 37, 40) | 11 | 11
  Day 41 (N= 32, 36) | 2 | 6
  Day 42 (N= 30, 35) | 7 | 6
  Day 43 (N= 25, 31) | 9 | 12
  Day 44 (N= 6, 7) | 1 | 1
  Day 45 (N= 3, 4) | 2 | 1
  Day 46 (N= 3, 2) | 1 | 1
  Day 47 (N= 1, 1) | 0 | 0
  Day 48 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 49 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 50 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 51 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 52 (N= 1, 1) | 0 | 0
  Day 53 (N= 1, 1) | 0 | 0
  Day 54 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 55 (N= 1, 1) | 0 | 0
  Day 56 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 57 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 58 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 59 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 60 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0

28. Secondary Outcome: Rehabilitation Parameter by Study Day- Number of Participants Who Were Able to Walk Without Assistance
Description: The number of participants responding affirmative in their rehabilitation diaries for each day
Time Frame: 60 days
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | FLOSEAL + Standard of Care (SoC) | Standard of Care (SoC)
Number analyzed (Participants) | 47 | 50
participants
  Day 1 (N= 47, 50) | 1 | 2
  Day 2 (N= 47, 50) | 1 | 1
  Day 3 (N= 46, 50) | 0 | 1
  Day 4 (N= 46, 48) | 0 | 3
  Day 5 (N= 42, 44) | 5 | 2
  Day 6 (N= 40, 42) | 7 | 4
  Day 7 (N= 40, 42) | 8 | 5
  Day 8 (N= 38, 42) | 6 | 4
  Day 9 (N= 37, 41) | 5 | 7
  Day 10 (N= 34, 40) | 5 | 6
  Day 11 (N= 36, 41) | 7 | 8
  Day 12 (N= 36, 39) | 8 | 10
  Day 13 (N= 38, 39) | 9 | 11
  Day 14 (N= 39, 39) | 10 | 11
  Day 15 (N= 40, 42) | 9 | 14
  Day 16 (N= 40, 41) | 10 | 13
  Day 17 (N= 38, 41) | 10 | 16
  Day 18 (N= 40, 41) | 10 | 16
  Day 19 (N= 41, 41) | 12 | 15
  Day 20 (N= 40, 40) | 14 | 15
  Day 21 (N= 39, 40) | 14 | 16
  Day 22 (N= 39, 41) | 15 | 16
  Day 23 (N= 39, 40) | 16 | 18
  Day 24 (N= 40, 39) | 16 | 18
  Day 25 (N= 39, 40) | 17 | 20
  Day 26 (N= 39, 39) | 18 | 18
  Day 27 (N= 39, 39) | 18 | 21
  Day 28 (N= 38, 39) | 19 | 22
  Day 29 (N= 38, 39) | 19 | 20
  Day 30 (N= 36, 40) | 20 | 26
  Day 31 (N= 37, 40) | 21 | 27
  Day 32 (N= 37, 40) | 23 | 25
  Day 33 (N= 38, 39) | 23 | 27
  Day 34 (N= 37, 39) | 23 | 27
  Day 35 (N= 38, 39) | 23 | 28
  Day 36 (N= 38, 40) | 22 | 29
  Day 37 (N= 36, 39) | 23 | 28
  Day 38 (N= 36, 41) | 24 | 30
  Day 39 (N= 36, 39) | 24 | 29
  Day 40 (N= 37, 40) | 25 | 30
  Day 41 (N= 32, 36) | 23 | 27
  Day 42 (N= 31, 35) | 22 | 26
  Day 43 (N= 25, 31) | 18 | 24
  Day 44 (N= 6, 8) | 5 | 5
  Day 45 (N= 3, 4) | 2 | 4
  Day 46 (N= 3, 2) | 2 | 2
  Day 47 (N= 1, 1) | 0 | 1
  Day 48 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 1
  Day 49 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 1
  Day 50 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 1
  Day 51 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 1
  Day 52 (N= 1, 1) | 0 | 1
  Day 53(N= 1, 1) | 0 | 1
  Day 54 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 1
  Day 55 (N= 1, 1) | 0 | 1
  Day 56 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 1
  Day 57 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 1
  Day 58 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 1
  Day 59 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 1
  Day 60 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 1

29. Secondary Outcome: Rehabilitation Parameter by Study Day- Number of Participants Who Were Using a Walker
Description: The number of participants responding affirmative in their rehabilitation diaries for each day
Time Frame: 60 days
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | FLOSEAL + Standard of Care (SoC) | Standard of Care (SoC)
Number analyzed (Participants) | 47 | 50
participants
  Day 1 (N= 47, 50) | 17 | 20
  Day 2 (N= 47, 50) | 39 | 41
  Day 3 (N= 46, 50) | 38 | 46
  Day 4 (N= 46, 48) | 38 | 44
  Day 5 (N= 42, 44) | 33 | 40
  Day 6 (N= 40, 42) | 34 | 38
  Day 7 (N= 40, 42) | 32 | 38
  Day 8 (N= 38, 42) | 31 | 36
  Day 9 (N= 37, 41) | 26 | 34
  Day 10 (N= 34, 40) | 23 | 33
  Day 11 (N= 36, 41) | 24 | 32
  Day 12 (N= 36, 39) | 24 | 27
  Day 13 (N= 38, 39) | 26 | 22
  Day 14 (N= 39, 39) | 23 | 21
  Day 15 (N= 40, 42) | 19 | 22
  Day 16 (N= 40, 41) | 19 | 23
  Day 17 (N= 38, 41) | 17 | 21
  Day 18 (N= 40, 41) | 17 | 22
  Day 19 (N= 41,41 ) | 20 | 20
  Day 20 (N= 40, 40) | 15 | 19
  Day 21 (N= 39, 40) | 15 | 18
  Day 22 (N= 39, 41) | 12 | 17
  Day 23 (N= 39, 40) | 12 | 16
  Day 24 (N= 40, 39) | 12 | 14
  Day 25 (N= 39, 40) | 8 | 11
  Day 26 (N= 39, 39) | 9 | 9
  Day 27 (N= 39, 39) | 8 | 7
  Day 28 (N= 38, 39) | 9 | 6
  Day 29 (N= 38, 39) | 8 | 7
  Day 30 (N= 36, 40) | 5 | 7
  Day 31 (N= 37, 40) | 5 | 6
  Day 32 (N= 37, 40) | 8 | 6
  Day 33 (N= 38, 39) | 6 | 5
  Day 34 (N= 37, 39) | 5 | 5
  Day 35 (N= 38, 39) | 6 | 7
  Day 36 (N= 38, 40) | 5 | 5
  Day 37 (N= 36, 39) | 3 | 2
  Day 38 (N= 36, 41) | 4 | 4
  Day 39 (N= 36, 39) | 3 | 3
  Day 40 (N= 37, 40) | 4 | 3
  Day 41 (N= 32, 36) | 2 | 4
  Day 42 (N= 31, 35) | 2 | 3
  Day 43 (N= 25, 31) | 1 | 2
  Day 44 (N= 6, 8) | 0 | 1
  Day 45 (N= 3, 4) | 0 | 0
  Day 46 (N= 3, 2) | 0 | 0
  Day 47 (N= 1, 1) | 0 | 0
  Day 48 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 49(N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 50 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 51 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 52 (N= 1, 1) | 1 | 0
  Day 53 (N= 1, 1) | 1 | 0
  Day 54 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 55 (N= 1, 1) | 1 | 0
  Day 56 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 57 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 58 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 59 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 60 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0

30. Secondary Outcome: Rehabilitation Parameter by Study Day- Number of Participants Who Were Using a Walking Cane
Description: The number of participants responding affirmative in their rehabilitation diaries for each day
Time Frame: 60 days
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | FLOSEAL + Standard of Care (SoC) | Standard of Care (SoC)
Number analyzed (Participants) | 47 | 50
participants
  Day 1 (N= 47, 50) | 1 | 0
  Day 2 (N= 47, 50) | 0 | 0
  Day 3 (N= 46, 50) | 2 | 0
  Day 4 (N= 46, 48) | 1 | 3
  Day 5 (N= 42, 44) | 4 | 3
  Day 6 (N= 40, 42) | 2 | 3
  Day 7 (N= 40, 42) | 2 | 4
  Day 8 (N= 38, 42) | 2 | 6
  Day 9 (N= 37, 41) | 5 | 5
  Day 10 (N= 34, 40) | 6 | 6
  Day 11 (N= 36, 41) | 9 | 7
  Day 12 (N= 36, 39) | 11 | 10
  Day 13 (N= 38, 39) | 12 | 14
  Day 14 (N= 39, 39) | 16 | 12
  Day 15 (N= 40, 42) | 18 | 14
  Day 16 (N= 40, 41) | 20 | 15
  Day 17 (N= 38, 41) | 19 | 17
  Day 18 (N= 40, 41) | 19 | 18
  Day 19 (N= 41, 41) | 18 | 19
  Day 20 (N= 40, 40) | 18 | 22
  Day 21 (N= 39, 40) | 17 | 18
  Day 22 (N= 39, 41) | 20 | 20
  Day 23 (N= 39, 40) | 20 | 18
  Day 24 (N= 40, 39) | 20 | 17
  Day 25 (N= 39, 40) | 19 | 19
  Day 26 (N= 39, 39) | 21 | 21
  Day 27 (N= 39, 39) | 18 | 20
  Day 28 (N= 38, 39) | 18 | 19
  Day 29 (N= 38, 39) | 17 | 19
  Day 30 (N= 36, 40) | 16 | 17
  Day 31 (N= 37, 40) | 17 | 18
  Day 32 (N= 37, 40) | 14 | 18
  Day 33 (N= 38, 39) | 15 | 15
  Day 34 (N= 37, 39) | 15 | 16
  Day 35 (N= 38, 39) | 14 | 13
  Day 36 (N= 38, 40) | 15 | 17
  Day 37 (N= 36, 39) | 13 | 15
  Day 38 (N= 36, 41) | 10 | 16
  Day 39 (N= 36, 39) | 13 | 14
  Day 40 (N= 37, 40) | 11 | 15
  Day 41 (N= 32, 36) | 9 | 11
  Day 42 (N= 31, 35) | 7 | 11
  Day 43 (N= 25, 31) | 7 | 9
  Day 44 (N= 6, 8) | 1 | 1
  Day 45 (N= 3, 4) | 1 | 0
  Day 46 (N= 3, 2) | 1 | 0
  Day 47 (N= 1, 1) | 1 | 1
  Day 48 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 49 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 50 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 51 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 52 (N= 1, 1) | 0 | 0
  Day 53 (N= 1, 1) | 0 | 0
  Day 54 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 55 (N= 1, 1) | 1 | 0
  Day 56 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 57 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 58 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 59 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 60 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0

31. Secondary Outcome: Rehabilitation Parameter by Study Day- Number of Participants Who Were Using a Wheelchair
Description: The number of participants responding affirmative in their rehabilitation diaries for each day
Time Frame: 60 days
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | FLOSEAL + Standard of Care (SoC) | Standard of Care (SoC)
Number analyzed (Participants) | 47 | 50
participants
  Day 1 (N= 47, 50) | 0 | 0
  Day 2 (N= 47, 50) | 1 | 1
  Day 3 (N= 46, 50) | 1 | 1
  Day 4 (N= 46, 48) | 2 | 1
  Day 5 (N= 42, 44) | 7 | 5
  Day 6 (N= 40, 42) | 5 | 3
  Day 7 (N= 40, 42) | 4 | 3
  Day 8 (N= 38, 42) | 6 | 5
  Day 9 (N= 37, 41) | 5 | 4
  Day 10 (N= 34, 40) | 4 | 3
  Day 11 (N= 36, 41) | 4 | 3
  Day 12 (N= 36, 39) | 3 | 2
  Day 13 (N= 38, 39) | 2 | 2
  Day 14 (N= 39, 39) | 3 | 2
  Day 15 (N= 40, 42) | 4 | 5
  Day 16 (N= 40, 41) | 4 | 3
  Day 17 (N= 38, 41) | 4 | 2
  Day 18 (N= 40, 41) | 3 | 2
  Day 19 (N= 41, 41) | 4 | 2
  Day 20 (N= 40, 40) | 3 | 1
  Day 21 (N= 39, 40) | 2 | 1
  Day 22 (N= 39, 41) | 1 | 1
  Day 23 (N= 39, 40) | 3 | 1
  Day 24 (N= 40, 39) | 2 | 1
  Day 25 (N= 39, 40) | 3 | 1
  Day 26 (N= 39, 39) | 1 | 1
  Day 27 (N= 39, 39) | 2 | 0
  Day 28 (N= 38, 39) | 2 | 0
  Day 29 (N= 38, 39) | 2 | 1
  Day 30 (N= 36, 40) | 2 | 1
  Day 31 (N= 37, 40) | 2 | 1
  Day 32 (N= 37, 40) | 1 | 0
  Day 33 (N= 38, 39) | 2 | 0
  Day 34 (N= 37, 39) | 1 | 0
  Day 35 (N= 38, 39) | 2 | 0
  Day 36 (N= 38, 40) | 2 | 0
  Day 37 (N= 36, 39) | 1 | 0
  Day 38 (N= 36, 41) | 1 | 0
  Day 39 (N= 36, 39) | 1 | 0
  Day 40 (N= 37, 40) | 0 | 0
  Day 41 (N= 32, 36) | 1 | 0
  Day 42 (N= 31, 35) | 0 | 0
  Day 43 (N= 25, 31) | 0 | 0
  Day 44 (N= 6,8 ) | 0 | 0
  Day 45 (N= 3, 4) | 0 | 0
  Day 46 (N= 3, 2) | 0 | 0
  Day 47 (N= 1, 1) | 0 | 0
  Day 48 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 49 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 50 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 51 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 52 (N= 1, 1) | 0 | 0
  Day 53(N= 1, 1) | 0 | 0
  Day 54 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 55 (N= 1, 1) | 0 | 0
  Day 56 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 57 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 58 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 59 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 60 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0

32. Secondary Outcome: Rehabilitation Parameter by Study Day- Number of Participants Who Were Using a Another Walking Device (Other Than a: Walker, Walking Cane, or Wheelchair)
Description: The number of participants responding affirmative in their rehabilitation diaries for each day
Time Frame: 60 days
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | FLOSEAL + Standard of Care (SoC) | Standard of Care (SoC)
Number analyzed (Participants) | 47 | 50
participants
  Day 1 (N= 47, 50) | 0 | 0
  Day 2 (N= 47, 50) | 1 | 0
  Day 3 (N= 46, 50) | 3 | 0
  Day 4 (N= 46, 48) | 4 | 1
  Day 5 (N= 42, 44) | 6 | 2
  Day 6 (N= 40, 42) | 4 | 2
  Day 7 (N= 40, 42) | 6 | 2
  Day 8 (N= 38, 42) | 5 | 2
  Day 9 (N= 37, 41) | 5 | 3
  Day 10 (N= 34, 40) | 7 | 3
  Day 11 (N= 36, 41) | 6 | 3
  Day 12 (N= 36, 39) | 6 | 3
  Day 13 (N= 38, 39) | 6 | 3
  Day 14 (N= 39, 39) | 4 | 3
  Day 15 (N= 40, 42) | 5 | 5
  Day 16 (N= 40, 41) | 4 | 3
  Day 17 (N= 38, 41) | 4 | 2
  Day 18 (N= 40, 41) | 4 | 2
  Day 19 (N= 41, 41) | 3 | 3
  Day 20 (N= 40, 40) | 2 | 2
  Day 21 (N= 39, 40) | 2 | 2
  Day 22 (N= 39, 41) | 2 | 2
  Day 23 (N= 39, 40) | 2 | 2
  Day 24 (N= 40, 39) | 4 | 3
  Day 25 (N= 39, 40) | 2 | 2
  Day 26 (N= 39, 39) | 2 | 2
  Day 27 (N= 39, 39) | 2 | 2
  Day 28 (N= 38, 39) | 1 | 1
  Day 29 (N= 38, 39) | 1 | 2
  Day 30 (N= 36, 40) | 1 | 1
  Day 31 (N= 37, 40) | 1 | 1
  Day 32 (N= 37, 40) | 1 | 1
  Day 33 (N= 38, 39) | 0 | 1
  Day 34 (N= 37, 39) | 0 | 1
  Day 35 (N= 38, 39) | 0 | 1
  Day 36 (N= 38, 40) | 0 | 0
  Day 37 (N= 36, 39) | 1 | 0
  Day 38 (N= 36, 41) | 0 | 1
  Day 39 (N= 36, 39) | 2 | 0
  Day 40 (N= 37, 40) | 0 | 0
  Day 41 (N= 32, 36) | 0 | 0
  Day 42 (N= 31, 35) | 0 | 0
  Day 43 (N= 25, 31) | 0 | 0
  Day 44 (N= 6, 8) | 0 | 0
  Day 45 (N= 3, 4) | 0 | 0
  Day 46 (N= 3, 2) | 0 | 0
  Day 47 (N= 1, 1) | 0 | 0
  Day 48 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 49 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 50 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 51 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 52 (N= 1, 1) | 0 | 0
  Day 53 (N= 1, 1) | 0 | 0
  Day 54 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 55 (N= 1, 1) | 0 | 0
  Day 56 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 57 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 58 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 59 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 60 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0

33. Secondary Outcome: Rehabilitation Parameter by Study Day- Number of Participants Who Cannot Get Out of Bed
Description: The number of participants responding affirmative in their rehabilitation diaries for each day
Time Frame: 60 days
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | FLOSEAL + Standard of Care (SoC) | Standard of Care (SoC)
Number analyzed (Participants) | 47 | 50
participants
  Day 1 (N= 47, 50) | 23 | 27
  Day 2 (N= 47, 50) | 4 | 5
  Day 3 (N= 46, 50) | 3 | 0
  Day 4 (N= 46, 48) | 2 | 0
  Day 5 (N= 42, 44) | 1 | 2
  Day 6 (N= 42, 42) | 1 | 0
  Day 7 (N= 40, 42) | 0 | 0
  Day 8 (N= 38, 42) | 0 | 0
  Day 9 (N= 37, 41) | 0 | 0
  Day 10 (N= 34, 40) | 1 | 0
  Day 11 (N= 36, 41) | 0 | 0
  Day 12 (N= 36, 39) | 0 | 0
  Day 13 (N= 38, 39) | 0 | 0
  Day 14 (N= 39, 39) | 0 | 0
  Day 15 (N= 40, 42) | 0 | 0
  Day 16 (N= 40, 41) | 0 | 0
  Day 17 (N= 38, 41) | 0 | 0
  Day 18 (N= 40, 41) | 0 | 0
  Day 19 (N= 41, 41) | 0 | 0
  Day 20 (N= 40, 40) | 0 | 0
  Day 21 (N= 39, 40) | 0 | 0
  Day 22 (N= 39, 41) | 0 | 0
  Day 23 (N= 39, 40) | 0 | 0
  Day 24 (N= 40, 39) | 0 | 0
  Day 25 (N= 39, 40) | 0 | 0
  Day 26 (N= 39, 39) | 0 | 0
  Day 27 (N= 39, 39) | 0 | 0
  Day 28 (N= 38, 39) | 0 | 0
  Day 29 (N= 38, 39) | 0 | 1
  Day 30 (N= 36, 40) | 0 | 0
  Day 31 (N= 37, 40) | 0 | 0
  Day 32 (N= 37, 40) | 0 | 0
  Day 33 (N= 38, 39) | 0 | 0
  Day 34 (N= 37, 39) | 0 | 0
  Day 35 (N= 38, 39) | 0 | 0
  Day 36 (N= 38, 40) | 0 | 0
  Day 37 (N= 36, 39) | 0 | 0
  Day 38 (N= 36, 41) | 0 | 0
  Day 39 (N= 36, 39) | 0 | 0
  Day 40 (N= 37, 40) | 0 | 0
  Day 41 (N= 32, 36) | 0 | 0
  Day 42 (N= 31, 35) | 0 | 0
  Day 43 (N= 25, 31) | 0 | 0
  Day 44 (N= 6, 8) | 0 | 0
  Day 45 (N= 3, 4) | 0 | 0
  Day 46 (N= 3, 2) | 0 | 0
  Day 47 (N= 1, 1) | 0 | 0
  Day 48 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 49 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 50 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 51 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 52 (N= 1, 1) | 0 | 0
  Day 53 (N= 1, 1) | 0 | 0
  Day 54 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 55 (N= 1, 1) | 0 | 0
  Day 56 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 57 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 58 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 59 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 60 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0

34. Secondary Outcome: Rehabilitation Parameter by Study Day- Number of Participants Who Had Someone Helping Them to Walk
Description: The number of participants responding affirmative in their rehabilitation diaries for each day
Time Frame: 60 days
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | FLOSEAL + Standard of Care (SoC) | Standard of Care (SoC)
Number analyzed (Participants) | 47 | 50
participants
  Day 1 (N= 47, 50) | 2 | 2
  Day 2 (N= 47, 50) | 13 | 12
  Day 3 (N= 46, 50) | 13 | 13
  Day 4 (N= 46, 48) | 10 | 12
  Day 5 (N= 42, 44) | 5 | 5
  Day 6 (N= 40, 42) | 5 | 5
  Day 7 (N= 40, 42) | 4 | 2
  Day 8 (N= 38, 42) | 5 | 3
  Day 9 (N= 37, 41) | 4 | 1
  Day 10 (N= 34, 40) | 0 | 1
  Day 11 (N= 36, 41) | 0 | 1
  Day 12 (N= 36, 39) | 0 | 1
  Day 13 (N= 38, 39) | 0 | 1
  Day 14 (N= 39, 39) | 0 | 1
  Day 15 (N= 40, 42) | 0 | 1
  Day 16 (N= 40, 41) | 0 | 1
  Day 17 (N= 38, 41) | 0 | 1
  Day 18 (N= 40, 41) | 0 | 1
  Day 19 (N= 41,41 ) | 0 | 1
  Day 20 (N= 40, 40) | 0 | 1
  Day 21 (N= 39, 40) | 0 | 1
  Day 22 (N= 39, 41) | 0 | 1
  Day 23 (N= 39, 40) | 0 | 1
  Day 24 (N= 40, 39) | 0 | 1
  Day 25 (N= 39, 40) | 0 | 1
  Day 26 (N= 39, 39) | 0 | 1
  Day 27 (N= 39, 39) | 0 | 1
  Day 28 (N= 38, 39) | 0 | 1
  Day 29 (N= 38, 39) | 0 | 1
  Day 30 (N= 36, 40) | 0 | 1
  Day 31 (N= 37, 40) | 0 | 0
  Day 32 (N= 37, 40) | 0 | 1
  Day 33 (N= 38, 39) | 0 | 1
  Day 34 (N= 37, 39) | 0 | 0
  Day 35 (N= 38, 39) | 0 | 1
  Day 36 (N= 38, 40) | 0 | 1
  Day 37 (N= 36, 39) | 0 | 1
  Day 38 (N= 36, 41) | 0 | 0
  Day 39 (N= 36, 39) | 0 | 0
  Day 40 (N= 37, 40) | 0 | 0
  Day 41 (N= 32, 36) | 0 | 0
  Day 42 (N= 31, 35) | 0 | 0
  Day 43 (N= 25, 31) | 0 | 0
  Day 44 (N= 6, 8) | 0 | 0
  Day 45 (N= 3, 4) | 0 | 0
  Day 46 (N= 3, 2) | 0 | 0
  Day 47 (N= 1, 1) | 0 | 0
  Day 48 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 49 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 50 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 51 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 52 (N= 1, 1) | 0 | 0
  Day 53 (N= 1, 1) | 0 | 0
  Day 54 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 55 (N= 1, 1) | 0 | 0
  Day 56 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 57 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 58 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 59 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0
  Day 60 (N= 0, 1) | NA — No participants provided a response/assessment to this parameter for this time point | 0

ADVERSE EVENTS:
Time Frame: Throughout the study period 1 year and 4 months
Description: The FLOSEAL + Standard of Care (SoC) arm/group includes the 12 Run-In participants.
  Run-In = The first participant who qualified for surgery at each site was treated with FLOSEAL + SoC to allow the investigator to familiarize with the study procedures and the use of FLOSEAL.
Arm/Group | FLOSEAL + Standard of Care (SoC) | Standard of Care (SoC)
Serious Adverse Events (participants affected / at risk) | 4/65 | 6/53
Other Adverse Events (participants affected / at risk) | 5/65 | 3/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FLOSEAL + Standard of Care (SoC) (N=65) | Standard of Care (SoC) (N=53)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CORONARY ARTERY BYPASS (Surgical and medical procedures) | 0 (0) | 1 (1)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL DISCHARGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FLOSEAL + Standard of Care (SoC) (N=65) | Standard of Care (SoC) (N=53)
Anxiety (Psychiatric disorders) | 1 (1) | 3 (3)
Hypotension (Vascular disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or 1 year after study completion. Baxter requires a review of results communications (e.g., for confidential information) ≥30 days prior to submission or communication. Baxter may request an additional delay of ≤60 days(e.g., for intellectual property protection)